CLINICAL TRIAL: NCT05119374
Title: Clinical Evaluation of the Capability of SenseGuard™ Non-invasive Wearable Device, to Detect Respiratory Changes, During Home Monitoring of Subjects With High Susceptibility for Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AECOPD)
Brief Title: Clinical Evaluation of SenseGuard™ to Detect Respiratory Changes, During Home Monitoring of Subjects With High Risk of AECOPD.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NanoVation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PD-CLN-003
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: All subjects will receive the Investigational device - SenseGuard for daily measurement of respiratory parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational SenseGuard Device (Experimental): All subjects use SenseGuard Device for twice daily monitoring of respiratory parameters.
  Interventions: Device: SenseGuard Investigational Device

INTERVENTIONS:
Device: SenseGuard Investigational Device — SG is a wireless, wearable medical device, which includes nano-based sensors. It can seamlessly measure patient's tidal breathing during daily activities. SG extracts series of critical respiratory parameters, including; Respiration Rate (RR), Inhalation and Exhalation duration and ratio (I/E), as well as novel biomarkers. SG parameters are applicable to evaluate COPD patients' condition, or for monitoring patients with other respiratory conditions.
  SG components are:
  * RSM (Respiratory Sensing Module): non-invasive module with sensors that can detect the exhaled humidity and condensation. The RSM is a non-sterile, disposable, single patient use.
  * ECU (Electronic Control Unit): a re-usable, wireless data acquisition and transmission unit. The ECU is connected to the RSM during the measurement and transmits the data via Bluetooth to the SG software.
  * SenseGuard™ Software: for data management, acquisition, processing, logging and presentation of the digital respiratory signals.

SUMMARY:
This is an observational, open labeled study. The study aims to evaluate the capability of SenseGuard™ (SG) non-invasive wearable device, to detect, post-hoc, early respiratory changes due to exacerbation by daily monitoring of subjects with COPD, at home.

Subjects with COPD, that were discharged following hospitalization due to AECOPD are most susceptible to experience another exacerbation during the first 6 months post admission. Hence, subjects that were discharged from the hospital due to AECOPD during the last 3 months are eligible to the study.

DETAILED DESCRIPTION:
During the study subject will be monitored daily for up to 6 months. Subject will perform 2 daily measurements of tidal breathing with SG, for 8 minutes each. Measurements are performed at the same time window every day; in the morning, before any treatment, and in the evening.

Monitoring will be continued during exacerbations and hospitalization if and when occurred.

Subject will complete a weekly online COPD symptoms assessment questionnaire, sent by email or a text massage.

Subject will report the clinical team about any increase of respiratory symptoms that may lead to exacerbation. Subject will get treatment for confirmed exacerbation according to the Standard of Care. Each case of symptoms and/or confirmed exacerbation will be documented in the CRF and reported to NanoVation team within 24 hours from onset. The daily data obtained by SG, prior to the exacerbation, will be analyzed to detect early respiratory change associated with this exacerbation. This information is critical for SG data interpretation and for the development of early alert for AECOPD.

NanoVation team will provide all subjects with the following: training to use SG, technical support in any case of a problem with the device and reminders to use the SG in case of reduced compliance.

Study will include 3 visits:

Visit 1 - Enrolment visit (Day 0): will be conducted during subject hospitalization or at discharge day, or by inviting eligible subjects to this visit (subjects who were hospitalized during the last 3 months due to AECOPD).

Enrolment of eligible subjects by the clinical team will include:

* Review of medical record and diagnosis.
* Evaluation of Inclusion/ exclusion criteria.
* Subject receives explanation about study.
* Subject signs the Informed Consent form (ICF).
* Subject performs baseline Spirometry test.
* Subject fills a baseline COPD symptoms assessment questionnaire (CSAQ).
* Next visits are scheduled.
* Subject receives the SG home kit
* Subject is trained for self-operation of SG measurement.
* Subject's data is documented in the CRF.

Visit 2- Follow up visit (at 3 months) Subject will have a routine clinical follow up 3 months after discharge and recruitment to the study. During this visit, subject will undergo a routine spirometry breathing test and complete a usability questionnaire evaluating the daily experience with SG measurement. All data will be documented in the CRF.

Visit 3- End of study visit (at 6 months) Subject will have a routine clinical follow up, Subject will undergo a routine spirometry breathing test and will complete a SG usability questionnaire. Subject will return the SG home kit and all data will be documented in the CRF.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18.
2. Diagnosed with COPD, 30%< FEV1 <80% predicated, or FEV1>80% and FEV1/FVC < 0.7
3. Discharged from the hospital during the last 3 months due to AECOPD.
4. Provision of signed and dated informed consent form.
5. Speak, read and understand either Hebrew, Arabic or English.
6. Able to understand study requirements and comply with study procedures.
7. Able to operate a tablet for SG measurement.

Exclusion Criteria:

1. Suffer from any physical or cognitive impairment that may affect subject's capability to operate the SG device properly.
2. Pregnant woman or nursing mother.
3. Severely ill with less than 12-month life expectancy
4. Suffering from serious uncontrolled medical conditions that may interfere with study requirements.
5. Participated in another clinical study during the study period, that may interrupt their participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Significant changes in SenseGuard device respiratory parameters (Ratio of Inhalation to exhalation time) can indicate for early exacerbation of COPD patient. | 6 months
  60% of confirmed COPD exacerbations can be detected in post-hoc analysis of changes in tidal breathing parameters measured by SenseGuard™ (significant change from baseline of Ratio of Inhalation to Exhalation time).

SECONDARY OUTCOMES:
Rate of retention and Compliance of COPD patients who use SG for home monitoring | 6 months
  At least 60% of subjects completed at least 1 month of home monitoring by SG and were compliant to the study protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Nazzal, Dr., Principal Investigator — Poria Medical Center, Israel; Yaniv Dotan, Dr., Principal Investigator — Rambam Health Campus, Haifa, Israel
Locations (6):
- Israel (6):
  - The Barzilai University Medical Center, Ashkelon
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Campus, Haifa
  - Nazareth Hospital E.M.M.S, Nazareth
  - Tel Aviv Medical Center, Tel Aviv
  - The Institute of Pulmonology Baruch Padeh Medical Center, Tiberias